CLINICAL TRIAL: NCT00765050
Title: A Prospective, Open, Non-randomized Phase I/II Study of Therapeutic Angiogenesis in Diabetic Patients With Critic Ischemia of Lower Limbs While Administering Positive CD133 Mobilized With G-CSF
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: PETHEMA Foundation, PETHEMA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-000693-20
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Patients With Critic Ischemia in Lower Limbs Who Are Administered With CD133+ Cells Mobilized by G-CSF
Keywords: Cellular therapy; CD133+
MeSH Terms: conditions — Macular Dystrophy, Retinal, 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD133+ cells (Experimental): CD133+ cells, obtained from peripheral blood in the treatment of diabetic patients with critic ischemia in lower limbs.
  Interventions: Biological: CD133+ cells transplant

INTERVENTIONS:
Biological: CD133+ cells transplant — intramuscular administration of CD133+ cells that have been mobilized from peripheral blood.

SUMMARY:
The primary objective is to analyze the safety and efficacy of CD133+ cells, obtained from peripheral blood in the treatment of diabetic patients with critic ischemia in lower limbs.

The secondary objectives are:

* To determine the safety of the intramuscular administration of CD133+ cells that have been mobilized from peripheral blood.
* To determine the CD133+ capacity to increase the re-vascularization at lower limbs in diabetic patients with critic ischemia in the lower limbs.
* To evaluate the patient global health condition using the notified results of the SF-36 questionnaires completed by patients

DETAILED DESCRIPTION:
A total of up to 20 diabetic patients with critic ischemia of lower limbs will be included in the study. Patients will be administered with CD133+ cells, that previously have been obtained of their peripheral blood after mobilization with G-CSF

The study is divided in three phases:

Pre-treatment (previous 4 weeks of CD133+ cells mobilization). Treatment (cells mobilization, CD133+ transplant, 24 hours after infusion visit, 4, 12 and 24 weeks after transplant visits) Follow-up (9 and 12 months after transplant visits)

ELIGIBILITY:
Inclusion Criteria:

* According to the investigator opinion, patient is able to carry out with all the clinical trial requirements
* Patient must volunteer sign the inform consent before any study specific test, that is not part of the common patient attention, is performed. Patient must know that he/she can abandon the study at any time with no damage to his/her posterior attention
* Age 18 to 75
* A diagnosis of chronic critic ischemia of the lower limbs
* Diabetes Mellitus active
* III or IV stages (Fontaine classification): resting pain, ulcer or minor gangrene with no major amputation
* General contraindication or local inoperability or refractory/progression after previous surgical treatment, according to the investigator criteria
* If female reproductive potential, negative pregnancy test

Exclusion Criteria:

* Pregnant or currently breast feeding women
* Acute myocardial infarction within the last 3 years
* Non re-vascular unstable angina pectoris
* History of ischemia stroke within the last 3 years
* Neoplasia at the time of inclusion or Chemotherapy or Radiotherapy treatment in the last 5 years
* Chronic renal insufficiency
* G-CSF contraindication
* A non well controlled serious concomitant disease
* History of serious thrombotic episodes within the past 3 years
* Patients who have received other investigational therapy within 30 days previous to the study inclusion
* Patients currently in other clinical trial or receiving any other investigational agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
analyze the safety and efficacy of CD133+ cells, obtained from peripheral blood in the treatment of diabetic patients with critic ischemia in lower limbs. | 12 months

SECONDARY OUTCOMES:
To determine the safety of the intramuscular administration of CD133+ cells that have been mobilized from peripheral blood | 2 months
To determine the CD133+ capacity to increase the re-vascularization at lower limbs in diabetic patients with critic ischemia in the lower limbs | 12 months
To evaluate the patient global health condition using the notified results of the SF-36 questionnaires completed by patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mª Consuelo Del Cañizo, Dr, Study Chair — Hospital Clínico de Salamanca
Locations (5):
- Spain (5):
  - Hospital Virgen de la Arrixaca, Murcia
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Clínico Universitario, Salamanca
  - Hospital Joan XIII de, Tarragona
  - Hospital Clínico Universitario, Valladolid

REFERENCES:
- [Background] Second European Consensus Document on chronic critical leg ischemia. Circulation. 1991 Nov;84(4 Suppl):IV1-26. No abstract available. PMID 1834364
- [Background] Mohler ER 3rd. Therapy insight: peripheral arterial disease and diabetes--from pathogenesis to treatment guidelines. Nat Clin Pract Cardiovasc Med. 2007 Mar;4(3):151-62. doi: 10.1038/ncpcardio0823. PMID 17330127
- [Background] Dormandy JA, Rutherford RB. Management of peripheral arterial disease (PAD). TASC Working Group. TransAtlantic Inter-Society Consensus (TASC). J Vasc Surg. 2000 Jan;31(1 Pt 2):S1-S296. No abstract available. PMID 10666287
- [Background] Perez Encinas M, Fernandez MA, Martin ML, Calvo MV, Gomez-Alonso A, Dominguez-Gil A, Lozano F. Multicriteria decision analysis for determining drug therapy for intermittent claudication. Methods Find Exp Clin Pharmacol. 1998 Jun;20(5):425-31. doi: 10.1358/mf.1998.20.5.485704. PMID 9701781
- [Background] Ramos M, Almazan A, Lozano F, Gomez-Alonso A. Phenol lumbar sympathectomy in severe arterial disease of the lower limbs: a hemodynamic study. Int Surg. 1983 Apr-Jun;68(2):127-30. PMID 6885290
- [Background] Almeida J, Bueno C, Alguero MC, Sanchez ML, Canizo MC, Fernandez ME, Vaquero JM, Laso FJ, Escribano L, San Miguel JF, Orfao A. Extensive characterization of the immunophenotype and pattern of cytokine production by distinct subpopulations of normal human peripheral blood MHC II+/lineage- cells. Clin Exp Immunol. 1999 Dec;118(3):392-401. doi: 10.1046/j.1365-2249.1999.01078.x. PMID 10594557
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Asahara T, Masuda H, Takahashi T, Kalka C, Pastore C, Silver M, Kearne M, Magner M, Isner JM. Bone marrow origin of endothelial progenitor cells responsible for postnatal vasculogenesis in physiological and pathological neovascularization. Circ Res. 1999 Aug 6;85(3):221-8. doi: 10.1161/01.res.85.3.221. PMID 10436164
- [Background] Asahara T, Takahashi T, Masuda H, Kalka C, Chen D, Iwaguro H, Inai Y, Silver M, Isner JM. VEGF contributes to postnatal neovascularization by mobilizing bone marrow-derived endothelial progenitor cells. EMBO J. 1999 Jul 15;18(14):3964-72. doi: 10.1093/emboj/18.14.3964. PMID 10406801
- [Background] Canizo MC, Lozano F, Gonzalez-Porras JR, Barros M, Lopez-Holgado N, Briz E, Sanchez-Guijo FM. Peripheral endothelial progenitor cells (CD133 +) for therapeutic vasculogenesis in a patient with critical limb ischemia. One year follow-up. Cytotherapy. 2007;9(1):99-102. doi: 10.1080/14653240601034708. PMID 17354105
- [Background] de Wynter EA, Buck D, Hart C, Heywood R, Coutinho LH, Clayton A, Rafferty JA, Burt D, Guenechea G, Bueren JA, Gagen D, Fairbairn LJ, Lord BI, Testa NG. CD34+AC133+ cells isolated from cord blood are highly enriched in long-term culture-initiating cells, NOD/SCID-repopulating cells and dendritic cell progenitors. Stem Cells. 1998;16(6):387-96. doi: 10.1002/stem.160387. PMID 9831864
- [Background] Durdu S, Akar AR, Arat M, Sancak T, Eren NT, Ozyurda U. Autologous bone-marrow mononuclear cell implantation for patients with Rutherford grade II-III thromboangiitis obliterans. J Vasc Surg. 2006 Oct;44(4):732-9. doi: 10.1016/j.jvs.2006.06.023. Epub 2006 Aug 22. PMID 16926085
- [Background] Fadini GP, Sartore S, Albiero M, Baesso I, Murphy E, Menegolo M, Grego F, Vigili de Kreutzenberg S, Tiengo A, Agostini C, Avogaro A. Number and function of endothelial progenitor cells as a marker of severity for diabetic vasculopathy. Arterioscler Thromb Vasc Biol. 2006 Sep;26(9):2140-6. doi: 10.1161/01.ATV.0000237750.44469.88. Epub 2006 Jul 20. PMID 16857948
- [Background] Flamme I, Risau W. Induction of vasculogenesis and hematopoiesis in vitro. Development. 1992 Oct;116(2):435-9. doi: 10.1242/dev.116.2.435. PMID 1286617
- [Background] Folkman J. Tumor angiogenesis: therapeutic implications. N Engl J Med. 1971 Nov 18;285(21):1182-6. doi: 10.1056/NEJM197111182852108. No abstract available. PMID 4938153
- [Background] Fukumoto Y, Miyamoto T, Okamura T, Gondo H, Iwasaki H, Horiuchi T, Yoshizawa S, Inaba S, Harada M, Niho Y. Angina pectoris occurring during granulocyte colony-stimulating factor-combined preparatory regimen for autologous peripheral blood stem cell transplantation in a patient with acute myelogenous leukaemia. Br J Haematol. 1997 Jun;97(3):666-8. doi: 10.1046/j.1365-2141.1997.842724.x. PMID 9207419
- [Background] Gehling UM, Ergun S, Schumacher U, Wagener C, Pantel K, Otte M, Schuch G, Schafhausen P, Mende T, Kilic N, Kluge K, Schafer B, Hossfeld DK, Fiedler W. In vitro differentiation of endothelial cells from AC133-positive progenitor cells. Blood. 2000 May 15;95(10):3106-12. PMID 10807776
- [Background] Gill M, Dias S, Hattori K, Rivera ML, Hicklin D, Witte L, Girardi L, Yurt R, Himel H, Rafii S. Vascular trauma induces rapid but transient mobilization of VEGFR2(+)AC133(+) endothelial precursor cells. Circ Res. 2001 Feb 2;88(2):167-74. doi: 10.1161/01.res.88.2.167. PMID 11157668
- [Background] Gordon PR, Leimig T, Babarin-Dorner A, Houston J, Holladay M, Mueller I, Geiger T, Handgretinger R. Large-scale isolation of CD133+ progenitor cells from G-CSF mobilized peripheral blood stem cells. Bone Marrow Transplant. 2003 Jan;31(1):17-22. doi: 10.1038/sj.bmt.1703792. PMID 12621502
- [Background] Isner JM, Walsh K, Symes J, Pieczek A, Takeshita S, Lowry J, Rossow S, Rosenfield K, Weir L, Brogi E, et al. Arterial gene therapy for therapeutic angiogenesis in patients with peripheral artery disease. Circulation. 1995 Jun 1;91(11):2687-92. doi: 10.1161/01.cir.91.11.2687. No abstract available. PMID 7538919
- [Background] Jackson KA, Majka SM, Wang H, Pocius J, Hartley CJ, Majesky MW, Entman ML, Michael LH, Hirschi KK, Goodell MA. Regeneration of ischemic cardiac muscle and vascular endothelium by adult stem cells. J Clin Invest. 2001 Jun;107(11):1395-402. doi: 10.1172/JCI12150. PMID 11390421
- [Background] Kajiguchi M, Kondo T, Izawa H, Kobayashi M, Yamamoto K, Shintani S, Numaguchi Y, Naoe T, Takamatsu J, Komori K, Murohara T. Safety and efficacy of autologous progenitor cell transplantation for therapeutic angiogenesis in patients with critical limb ischemia. Circ J. 2007 Feb;71(2):196-201. doi: 10.1253/circj.71.196. PMID 17251666
- [Background] Kalka C, Masuda H, Takahashi T, Gordon R, Tepper O, Gravereaux E, Pieczek A, Iwaguro H, Hayashi SI, Isner JM, Asahara T. Vascular endothelial growth factor(165) gene transfer augments circulating endothelial progenitor cells in human subjects. Circ Res. 2000 Jun 23;86(12):1198-202. doi: 10.1161/01.res.86.12.1198. PMID 10864908
- [Background] Kawachi Y, Watanabe A, Uchida T, Yoshizawa K, Kurooka N, Setsu K. Acute arterial thrombosis due to platelet aggregation in a patient receiving granulocyte colony-stimulating factor. Br J Haematol. 1996 Aug;94(2):413-6. doi: 10.1046/j.1365-2141.1996.d01-1807.x. PMID 8759907
- [Background] Kalka C, Masuda H, Takahashi T, Kalka-Moll WM, Silver M, Kearney M, Li T, Isner JM, Asahara T. Transplantation of ex vivo expanded endothelial progenitor cells for therapeutic neovascularization. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3422-7. doi: 10.1073/pnas.97.7.3422. PMID 10725398
- [Background] Kocher AA, Schuster MD, Szabolcs MJ, Takuma S, Burkhoff D, Wang J, Homma S, Edwards NM, Itescu S. Neovascularization of ischemic myocardium by human bone-marrow-derived angioblasts prevents cardiomyocyte apoptosis, reduces remodeling and improves cardiac function. Nat Med. 2001 Apr;7(4):430-6. doi: 10.1038/86498. PMID 11283669
- [Background] Kolvenbach R, Kreissig C, Ludwig E, Cagiannos C. Stem cell use in critical limb ischemia. J Cardiovasc Surg (Torino). 2007 Feb;48(1):39-44. PMID 17308520
- [Background] Lang P, Bader P, Schumm M, Feuchtinger T, Einsele H, Fuhrer M, Weinstock C, Handgretinger R, Kuci S, Martin D, Niethammer D, Greil J. Transplantation of a combination of CD133+ and CD34+ selected progenitor cells from alternative donors. Br J Haematol. 2004 Jan;124(1):72-9. doi: 10.1046/j.1365-2141.2003.04747.x. PMID 14675410
- [Background] Luttun A, Carmeliet G, Carmeliet P. Vascular progenitors: from biology to treatment. Trends Cardiovasc Med. 2002 Feb;12(2):88-96. doi: 10.1016/s1050-1738(01)00152-9. PMID 11852257
- [Background] Murayama T, Tepper OM, Silver M, Ma H, Losordo DW, Isner JM, Asahara T, Kalka C. Determination of bone marrow-derived endothelial progenitor cell significance in angiogenic growth factor-induced neovascularization in vivo. Exp Hematol. 2002 Aug;30(8):967-72. doi: 10.1016/s0301-472x(02)00867-6. PMID 12160849
- [Background] Zhang HK, Li M, Feng H. [Autologous transplantation of peripheral blood stem cell in treatment of critical limb ischemia]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2007 Jul;36(4):360-3. doi: 10.3785/j.issn.1008-9292.2007.04.009. Chinese. PMID 17717827
- [Background] Orlic D, Kajstura J, Chimenti S, Jakoniuk I, Anderson SM, Li B, Pickel J, McKay R, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Bone marrow cells regenerate infarcted myocardium. Nature. 2001 Apr 5;410(6829):701-5. doi: 10.1038/35070587. PMID 11287958
- [Background] Orlic D, Kajstura J, Chimenti S, Limana F, Jakoniuk I, Quaini F, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Mobilized bone marrow cells repair the infarcted heart, improving function and survival. Proc Natl Acad Sci U S A. 2001 Aug 28;98(18):10344-9. doi: 10.1073/pnas.181177898. Epub 2001 Aug 14. PMID 11504914
- [Background] Peichev M, Naiyer AJ, Pereira D, Zhu Z, Lane WJ, Williams M, Oz MC, Hicklin DJ, Witte L, Moore MA, Rafii S. Expression of VEGFR-2 and AC133 by circulating human CD34(+) cells identifies a population of functional endothelial precursors. Blood. 2000 Feb 1;95(3):952-8. PMID 10648408
- [Background] Quirici N, Soligo D, Caneva L, Servida F, Bossolasco P, Deliliers GL. Differentiation and expansion of endothelial cells from human bone marrow CD133(+) cells. Br J Haematol. 2001 Oct;115(1):186-94. doi: 10.1046/j.1365-2141.2001.03077.x. PMID 11722432
- [Background] Risau W, Sariola H, Zerwes HG, Sasse J, Ekblom P, Kemler R, Doetschman T. Vasculogenesis and angiogenesis in embryonic-stem-cell-derived embryoid bodies. Development. 1988 Mar;102(3):471-8. doi: 10.1242/dev.102.3.471. PMID 2460305
- [Background] Simons M, Bonow RO, Chronos NA, Cohen DJ, Giordano FJ, Hammond HK, Laham RJ, Li W, Pike M, Sellke FW, Stegmann TJ, Udelson JE, Rosengart TK. Clinical trials in coronary angiogenesis: issues, problems, consensus: An expert panel summary. Circulation. 2000 Sep 12;102(11):E73-86. doi: 10.1161/01.cir.102.11.e73. PMID 10982554
- [Background] Stamm C, Westphal B, Kleine HD, Petzsch M, Kittner C, Klinge H, Schumichen C, Nienaber CA, Freund M, Steinhoff G. Autologous bone-marrow stem-cell transplantation for myocardial regeneration. Lancet. 2003 Jan 4;361(9351):45-6. doi: 10.1016/S0140-6736(03)12110-1. PMID 12517467
- [Background] Takahashi T, Kalka C, Masuda H, Chen D, Silver M, Kearney M, Magner M, Isner JM, Asahara T. Ischemia- and cytokine-induced mobilization of bone marrow-derived endothelial progenitor cells for neovascularization. Nat Med. 1999 Apr;5(4):434-8. doi: 10.1038/7434. PMID 10202935
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Background] Toma C, Pittenger MF, Cahill KS, Byrne BJ, Kessler PD. Human mesenchymal stem cells differentiate to a cardiomyocyte phenotype in the adult murine heart. Circulation. 2002 Jan 1;105(1):93-8. doi: 10.1161/hc0102.101442. PMID 11772882
- [Background] Tse HF, Kwong YL, Chan JK, Lo G, Ho CL, Lau CP. Angiogenesis in ischaemic myocardium by intramyocardial autologous bone marrow mononuclear cell implantation. Lancet. 2003 Jan 4;361(9351):47-9. doi: 10.1016/S0140-6736(03)12111-3. PMID 12517468
- [Background] Weiss MJ, Orkin SH. In vitro differentiation of murine embryonic stem cells. New approaches to old problems. J Clin Invest. 1996 Feb 1;97(3):591-5. doi: 10.1172/JCI118454. No abstract available. PMID 8609212
- See also: Spanish association of Haematology — http://www.aehh.org